CLINICAL TRIAL: NCT06449729
Title: Endocrine Determinants of Renal Function in Patients With Hypoparathyroidism on Conventional Treatment: a Cross-sectional Study
Brief Title: Endocrine Determinants of Renal Function in Patients With Hypoparathyroidism
Acronym: ENDORSE
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Andrea Giustina, Prorector and Head of Endocrinology, IRCCS San Raffaele
Other Study IDs: BP 11006333
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-03

CONDITIONS: Hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sample and urine collection — Blood sample and urine collection as per clinical practice

SUMMARY:
Endocrine determinants of renal function in patients with hypoparathyroidism on conventional treatment: a cross-sectional study (ENDORSE)

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* diagnosis of chronic (≥ 1 year) post-surgical and autoimmune hypoparathyroidism, as established with undetectable or insufficient PTH concentration in relation to the presence of hypocalcemia
* patients being treated with calcitriol or alfacalcidiol
* patients able to sign the written informed consent

Exclusion Criteria:

* pregnancy
* severe renal failure requiring dialysis treatment
* macroproteinuria
* use of antihypertensive drugs such as thiazides, ACE inhibitors, sartans, beta and alpha blockers, and antialdosterone drugs
* pazients affected by diabetes mellitus- insulin-treated

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with hypoparathyroidism being treated with calcitriol or alfacalcidiol.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
The rate of renal failure and altered PTH-related renal active hormonal axis in patients with hypoparathyroidism | 12 months
  Evaluation of the prevalence of renal failure and altered PTH-related renal active hormonal axis in patients with hypoparathyroidism (hypoPTH) in conventional treatment with calcium and vitamin D

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea Giustina, Milan, Italy